CLINICAL TRIAL: NCT04947280
Title: Single Arm Phase II Study of Fractionated Stereotatic Radiation Therapy (FSRT) for Bone Metastases in Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC012
Record Dates: First submitted 2021-04-08; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-04

CONDITIONS: Bone Metastases; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fractionated Stereotatic Radiation Therapy (Experimental)
  Interventions: Radiation: Fractionated Stereotatic Radiation Therapy

INTERVENTIONS:
Radiation: Fractionated Stereotatic Radiation Therapy — Participants prescribed to receive 9 Gy x 3 or 10 Gy x3 image-guided fractionated stereotatic radiation therapy.
  Other Names: Stereotatic Fractionated Radiation

SUMMARY:
Fractionated stereotatic radiation therapy (FSRT) that very precisely delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. The purpose of this study is to find out if FSRT is safe and effective in the treatment of metastatic spinal tumors of breast cancer.

DETAILED DESCRIPTION:
Eligible breast cancer patients with bone metastases will be treated with FSRT. 9-10 Gy x 3Fx or 6-7 Gy x 5Fx image-guided fractionated stereotatic radiation therapy will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of invasive breast cancer
2. Signed informed consent
3. Bone metastases (confirmed by MRI within 4 weeks of enrollment).
4. Paraosseous soft tissue ≤ 5cm. The tumour could involve the vertebral column, but did not have to, nor did it need to enter the spinal canal.
5. KPS ≥ 40 or ECOG 0-2.
6. The tumor is at least 2 mm away from the spinal cord. If the tumor is closer than 2 mm, surgical resection is required prior to FSRT or the total prescription dose of spinal cord is strictly limited.
7. Failure of previous conventional external beam radiotherapy or surgery, residual tumor after surgery, medical inoperability, and refusal to undergo surgery.
8. A maximum of three distinct noncontiguous spinal metastases per patient was allowed, and each of the separate sites may have involvement of 2 contiguous vertebral bodies.
9. Patients have sufficient bone marrow reserve and liver and kidney function: neutrophil count ≥ 1500 cells / mm3; platelet count ≥ 70000 / mm3; hemoglobin (Hgb) ≥ 8.0 g / dl; if there is liver metastasis, AST and ALT < 3x ULN
10. The interval between systemic chemotherapy is more than 2 weeks, and the side effects recovery from previous treatment ≤ grade 1
11. Patients receiving bisphosphonates, endocrine or targeted therapy at the same time were not included

Exclusion Criteria:

1. Patients with mechanically unstable spine or epidural spinal cord compression were excluded; however, patients with previously documented spinal cord compression that had been decompressed and stabilized were eligible. Patients with > 50% loss of vertebral body height were excluded.
2. Patients in whom a delay in initiating treatment might have adversely affected neurological outcome.
3. Patients with a pacemaker, unable to undergo MR imaging and unable to lie flat for at least 30 minutes.
4. Patients who had a history of previous radiotherapy to the spine at the current level of interest.
5. Patients who had received prior external-beam irradiation to the spine within 3 months of registration.
6. Patients who had received systemic radiotherapy (Strontium-89) within 30 days of starting protocol treatment.
7. Patients who had received chemotherapy within 2 weeks of starting protocol treatment.
8. Patients who are unwilling or unable to receive regular follow-up.
9. The patients judged by the researchers who could not be included in some special cases.
10. Serious complications: cardiovascular disease, end-stage renal disease, serious liver disease, infection, et al.
11. Pregnant women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Local Control Rate | 3 years
  Determine the local control rate of FSRT in patients with bone metastasis of breast cancer

SECONDARY OUTCOMES:
Pain Control | 3 years
  Evaluate whether FSRT improves pain control as measured by Brief Pain Inventory (BPI) after FSRT in patients with spinal metastasis of breast cancer
Overall Survival | 3 years
  Time from the date of informed consent until to the date of death, regardless of the cause of death
Progression Free Survival | 3 years
  Time from the date of radiotherapy to the investigator-determined date of progression or death due to any cause, whichever occurs first
Quality of Life | 3 years
  Evaluate the quality of life according to EORTC QLQ-BM22
Vertebral Fracture and Radiation Myelitis | 3 years
  Determine the incidence of bone fracture and radiation myelitis

CONTACTS AND LOCATIONS:
Overall Officials: Zhaozhi Yang, MD, Ph.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China